CLINICAL TRIAL: NCT03159273
Title: Dietary Supplementation of Nitrate by Beetroot Juice to Boost Immunity, Mood, Cardiovascular Function During Academic Stress
Brief Title: Nitrate Supplementation During Final Examination Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Thomas Ritz, Professor, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014_012_RITT
Record Dates: First submitted 2015-11-11; First posted 2017-05-18 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Airway Disease
Keywords: Dietary nitrate supplementation; Cold symptoms; Stress; Immunity; Exhaled nitric oxide; Lung function; Cardiovascular activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beetroot Juice Group (Experimental): Subjects in this group are given 7 daily doses of a dietary nitrate supplement (Beet-it Sport beetroot juice shots) and asked to drink one dose daily during the week of their final academic examinations of that term in college.
  Interventions: Dietary Supplement: Beetroot Juice Group
- Control (No Intervention): Subjects in this group are not given a dietary nitrate supplement but are assessed at the same time points as those in the experimental group.

INTERVENTIONS:
Dietary Supplement: Beetroot Juice Group — Beetroot juice drink- 7 daily doses (70 ml, containing 0.4-0.5 mg nitrate) taken over a week
  Other Names: Beet-It Sport Beet Juice Shot
  Arms: Beetroot Juice Group

SUMMARY:
The purpose of the present study is to explore the effects of a dietary nitrate supplement on immunity, mood, cardiovascular activity, and lung function during and following final exam stress in both healthy and asthmatic individuals.

DETAILED DESCRIPTION:
Past research has demonstrated significant changes in immune response and airway inflammation during times of stress. Specifically, significant decreases in the fraction of exhaled nitric oxide (FeNO) in both healthy and asthmatic undergraduate students have been found during times of final exam stress. Additionally, research suggests that dietary supplementation of nitric oxide may have beneficial cardiovascular effects which may offset the physiological consequences of stress.

This research study explores the effects of a dietary supplement on immunity, mood, cardiovascular and respiratory function during and following final exam stress. In this study, investigators monitor changes in respiratory infection incidence, airway nitric oxide, mood, blood pressure, and lung function in students with and without asthma during the time of final exams and a comparable time of low stress during the term. There are three assessments in the laboratory, as well as two additional brief questionnaires on separate days. During the final exam period, half of the participants are randomly assigned to the experimental group which is provided with a dietary supplement (beetroot juice drink) of which they are asked to take one dose every day in the morning for seven days. The three assessments periods include two during the week of final exams and one during a period of low stress scheduled up to two weeks to two months before that time. For the final exam period, the first of the two sessions takes place on the day before the second of these exams, and the second assessment takes place on a subsequent day after second exam. A follow-up assessment of cold symptoms takes place online 7 days after the final exam period.

ELIGIBILITY:
Inclusion Criteria:

* Lung healthy or physician diagnosis of asthma
* Undergraduate student with at least 3 final examinations

Exclusion Criteria:

* Current smoker
* History of seizures
* History of stroke
* History of heart attack or heart disease
* History of thyroid problems
* History of head injury or neurological disorder
* Diabetes
* Any kind of lung disease (other than asthma)
* Corticosteroids within the past month
* Antibiotics within the past month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Cold Symptoms | Non-stress assessment 2 weeks to 2 months before final exams, 2 assessments during the week of final exams (once the day before participants' 2nd final exam, and second on a day between 2nd and last exam); and 1 week post-exams
  Changes in participant-reported cold symptoms

SECONDARY OUTCOMES:
Change in Fraction of Exhaled Nitric Oxide (FeNO) | Non-stress assessment 2 weeks to 2 months before final exams, 2 assessments during the week of final exams (once the day before participants' 2nd final exam, and second on a day between 2nd and last exam);
  Changes in participant's measured level of nitric oxide in exhaled air
Change in Blood Pressure | Non-stress assessment 2 weeks to 2 months before final exams, 2 assessments during the week of final exams (once the day before participants' 2nd final exam, and second on a day between 2nd and last exam);
  Change in participant's measured systolic and diastolic blood pressure
Change in Forced Expiratory Volume in 1 second (FEV1) | Non-stress assessment 2 weeks to 2 months before final exams, 2 assessments during the week of final exams (once the day before participants' 2nd final exam, and second on a day between 2nd and last exam);
  Change in participant's measured FEV1 using a handheld spirometer
Change in Peak Expiratory Flow (PEF) | Non-stress assessment 2 weeks to 2 months before final exams, 2 assessments during the week of final exams (once the day before participants' 2nd final exam, and second on a day between 2nd and last exam);
  Change in participant's measured PEF using a handheld spirometer
Change in Negative Affect | Non-stress assessment 2 weeks to 2 months before final exams, 2 assessments during the week of final exams (once the day before participants' 2nd final exam, and second on a day between 2nd and last exam);
  PANAS negative affect scale

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ritz, Ph.D., Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

REFERENCES:
- [Derived] Ritz T, Werchan CA, Kroll JL, Rosenfield D. Beetroot juice supplementation for the prevention of cold symptoms associated with stress: A proof-of-concept study. Physiol Behav. 2019 Apr 1;202:45-51. doi: 10.1016/j.physbeh.2019.01.015. Epub 2019 Jan 22. PMID 30682333